CLINICAL TRIAL: NCT00191139
Title: A Randomized Study of Gemcitabine Plus Docetaxel After Cisplatin, Etoposide and Radiation Therapy in Stage III Unresectable NSCLC
Brief Title: Gemcitabine or Gemcitabine Plus Docetaxel After Cisplatin, Etoposide and Radiation in Non Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4697; B9E-US-S182 (Other: Eli Lilly and Company); NCT00074217 (obsolete NCT alias)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2009-12-25 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Docetaxel; Cisplatin; Etoposide; etoposide phosphate; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gemcitabine (Experimental)
  Interventions: Drug: gemcitabine; Drug: cisplatin; Drug: etoposide; Radiation: radiation therapy
- Gemcitabine plus Docetaxel (Experimental)
  Interventions: Drug: gemcitabine; Drug: docetaxel; Drug: cisplatin; Drug: etoposide; Radiation: radiation therapy

INTERVENTIONS:
Drug: gemcitabine — After induction chemotherapy, radiation therapy and 10 weeks with no disease progression, randomized consolidation treatment begins. In both treatment arms, gemcitabine 1000 milligrams per meter squared (mg/m2), is administered intravenously (IV), on days 1 and 8 of every 21-day cycle for 3 cycles.
  Other Names: LY188011; Gemzar
Drug: docetaxel — Following cisplatin-etoposide induction chemotherapy, radiation therapy and 10 weeks with no disease progression, randomized consolidation treatment begins. In this treatment arm, docetaxel 75 mg/m2, is administered IV on day 1 of each 21-day cycle for 3 cycles. Docetaxel is given after gemcitabine.
  Other Names: Taxotere
  Arms: Gemcitabine plus Docetaxel
Drug: cisplatin — As part of induction chemotherapy, cisplatin is given 50 mg/m2, IV, day 1, 8, 29 and 36 (spans 2 cycles)
  Other Names: Platinol; Platinol-AQ; CDDP
Drug: etoposide — As part of induction chemotherapy, etoposide is given 50 mg/m2, IV, days 1-5 and 29-33 (spans 2 cycles)
  Other Names: Toposar®; VePesid®; Etopophos®; VP-16; Etoposide phosphate
Radiation: radiation therapy — In conjunction with induction chemotherapy, radiation therapy is administered at a dose of 200 centi Gray (cGy) per day, Monday through Friday for 6 weeks

SUMMARY:
To assess the 2 year survival of patients with Stage III unresectable non-small cell lung cancer receiving consolidation gemcitabine or gemcitabine plus docetaxel following concurrent chemotherapy and radiation.

ELIGIBILITY:
Inclusion Criteria:

* histologic or cytologic proof of single primary non-small cell lung cancer
* No prior chemotherapy or radiation therapy
* no prior malignancy

Exclusion Criteria:

* pregnancy or breastfeeding
* serious concomitant systemic disorder
* unintentional weight loss greater than 10%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2003-03; Primary Completion 2008-11 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (15):
- United States (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, South Bend, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Kalamazoo, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Kansas City, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Memphis, Tennessee
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Rosario, Argentina
- China (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Chengdu
- South Korea (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Suwon

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine: Consolidation Treatment: gemcitabine 1000 milligrams per meter squared (mg/m2), is administered intravenously (IV), on days 1 and 8 of every 21-day cycle for 3 cycles
- Gemcitabine Plus Docetaxel: Consolidation Treatment: gemcitabine 1000 milligrams per meter squared (mg/m2), is administered intravenously (IV), on days 1 and 8 of every 21-day cycle for 3 cycles; docetaxel 75 mg/m2, is administered IV on day 1 of each 21-day cycle for 3 cycles. Docetaxel is given after gemcitabine.
Period: Overall Study
Arm/Group | Gemcitabine | Gemcitabine Plus Docetaxel
Started | 32 | 32
Completed | 27 | 20
Not Completed | 5 | 12
Not completed — Adverse Event | 2 | 6
Not completed — Death | 2 | 0
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Disease Progression | 0 | 1
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gemcitabine | Gemcitabine Plus Docetaxel | Total
Number analyzed (Participants) | 32 | 32 | 64
Age Continuous [Median (Standard Deviation); unit: years] | 59.5 (7.31) | 59.5 (9.61) | 59.5 (8.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 27 | 26 | 53
Race/Ethnicity, Customized [Number; unit: participants] — breakdown of participants by ethnic origin
  participants
    Caucasian | 18 | 19 | 37
    Black | 1 | 2 | 3
    Asian | 13 | 10 | 23
    Hispanic | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 18 | 20 | 38
  Argentina | 1 | 2 | 3
  China | 10 | 7 | 17
  Korea, Republic of | 3 | 3 | 6
Eastern Oncology Cooperative Group (ECOG) Performance Status [Number; unit: units on a scale] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  units on a scale
    0 - Fully Active | 12 | 14 | 26
    1 - Ambulatory, Restricted Strenuous Activity | 19 | 18 | 37
    2 - Ambulatory, No Work Activities | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: 2-Year Survival
Description: Percentage of participants alive at 2 years.
Time Frame: 2 years
Population: Intention to treat (ITT) population
Measure: Number; unit: percentage of participants
Arm/Group | Gemcitabine | Gemcitabine Plus Docetaxel
Number analyzed (Participants) | 32 | 32
percentage of participants | 40.6 | 55.7
Statistical Analysis 1: Comparison: Gemcitabine; Test type: Superiority or Other; normal approximation; Count the number of surviving participants at each time interval to get survival rates; survival rate = 40.6, 95% CI [23.8 to 56.8]
Statistical Analysis 2: Comparison: Gemcitabine Plus Docetaxel; Test type: Superiority or Other; normal approximation; Count the number of surviving participants at each time interval to get survival rates; survival rate = 55.7, 95% CI [36.8 to 70.9]

2. Secondary Outcome: Number of Patients With Overall Tumor Response
Description: Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria: Complete Response (CR)=disappearance of all target lesions; Partial Response (PR) =30% decrease in sum of longest diameter of target lesions; Progressive Disease (PD) =20% increase in sum of longest diameter of target lesions; Stable Disease (SD)=small changes that do not meet above criteria. The total number of CRs plus PRs equals overall response rate (ORR).
Time Frame: randomization and every 3 months up to 2 years of post-study followup
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Gemcitabine | Gemcitabine Plus Docetaxel
Number analyzed (Participants) | 32 | 32
participants | 24 | 27
Statistical Analysis 1: Comparison: Gemcitabine; Test type: Superiority or Other; normal approximation; Response Rate = 75, 95% CI [56.6 to 88.5]
Statistical Analysis 2: Comparison: Gemcitabine Plus Docetaxel; Test type: Superiority or Other; Normal approximation; Response rate = 84.4, 95% CI [67.2 to 94.7]

3. Secondary Outcome: Progression-Free Survival
Description: Defined as the time from randomization into consolidation treatment to the first date of documented disease progression or death. Progression-free survival time was censored at the date of the last follow-up visit at which disease was assessed for patients who were still alive and who had not progressed.
Time Frame: baseline to measured progressive disease up to 2057 days
Population: ITT population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Gemcitabine | Gemcitabine Plus Docetaxel
Number analyzed (Participants) | 32 | 32
days | 162.5 [82.0 to 239.0] | 408.0 [141.0 to 708.0]
Statistical Analysis 1: Comparison: Gemcitabine vs Gemcitabine Plus Docetaxel; Test type: Superiority or Other; p = 0.08, Log Rank

4. Secondary Outcome: Overall Survival
Description: Overall survival is the duration from enrollment to death from any cause. For patients who are alive, overall survival is censored at the last contact.
Time Frame: baseline to date of death from any cause up to 2057 days
Population: ITT population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Gemcitabine | Gemcitabine Plus Docetaxel
Number analyzed (Participants) | 32 | 32
days | 492.5 [299.0 to 1034.0] | 899.0 [498.0 to 1583.0]
Statistical Analysis 1: Comparison: Gemcitabine vs Gemcitabine Plus Docetaxel; Test type: Superiority or Other; p = 0.38, Log Rank

5. Secondary Outcome: Lung Cancer Symptom Scale (LCSS) Assessment Post-randomization
Description: LCSS measures physical & functional dimensions. The patient scale contains 9 items, 3 summation & 6 symptom items. Each item is marked on a visual analog scale (0=low; 100=high). The mean of the 6 symptoms is used to calculate the average symptom burden index (ASBI). Improved=mean ASBI assessments from any 2 consecutive improved post-randomization assessments was at least 0.5 standard deviation (SD) below pre-randomization ASBI; worse=mean ASBI from any 2 consecutive post-randomization assessments was at least 0.5 SD above pre-randomization ASBI; stable=criteria for improved/worse not met.
Time Frame: baseline to 3 months after last dose of study treatment (three 21-day cycles)
Population: as-treated population
Measure: Number; unit: participants
Arm/Group | Gemcitabine | Gemcitabine Plus Docetaxel
Number analyzed (Participants) | 32 | 32
participants
  Improvement | 8 | 5
  Stable | 10 | 9
  Worse | 2 | 8

ADVERSE EVENTS:
Arm/Group | Gemcitabine | Gemcitabine Plus Docetaxel
Serious Adverse Events (participants affected / at risk) | 13/32 | 18/32
Other Adverse Events (participants affected / at risk) | 32/32 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine (N=32) | Gemcitabine Plus Docetaxel (N=32)
Anaemia NOS (Blood and lymphatic system disorders) | 0 (0) | 4 (8)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Leukopenia NOS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 2 (6)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure NOS (Cardiac disorders) | 1 (1) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Oesophagitis NOS (Gastrointestinal disorders) | 1 (2) | 2 (3)
Vomiting NOS (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (2)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death NOS (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (2) | 2 (2)
Candidal infection NOS (Infections and infestations) | 0 (0) | 1 (1)
Lung infection NOS (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia NOS (Infections and infestations) | 4 (5) | 5 (5)
Sepsis NOS (Infections and infestations) | 0 (0) | 1 (1)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Convulsions NOS (Nervous system disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Face oedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine (N=32) | Gemcitabine Plus Docetaxel (N=32)
Anaemia NOS (Blood and lymphatic system disorders) | 18 (26) | 24 (63)
Erythropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Granulocytopenia (Blood and lymphatic system disorders) | 1 (2) | 2 (4)
Leukopenia NOS (Blood and lymphatic system disorders) | 12 (41) | 13 (41)
Lymphopenia (Blood and lymphatic system disorders) | 4 (6) | 3 (6)
Neutropenia (Blood and lymphatic system disorders) | 19 (93) | 23 (73)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (27) | 13 (33)
Tachycardia NOS (Cardiac disorders) | 7 (8) | 5 (5)
Tinnitus (Ear and labyrinth disorders) | 5 (5) | 3 (3)
Vision blurred (Eye disorders) | 1 (1) | 3 (3)
Abdominal pain NOS (Gastrointestinal disorders) | 2 (2) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 4 (5)
Constipation (Gastrointestinal disorders) | 13 (16) | 14 (25)
Diarrhoea NOS (Gastrointestinal disorders) | 9 (15) | 16 (22)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 9 (13)
Dysphagia (Gastrointestinal disorders) | 11 (15) | 13 (19)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (2)
Nausea (Gastrointestinal disorders) | 23 (54) | 28 (62)
Odynophagia (Gastrointestinal disorders) | 3 (5) | 2 (3)
Oesophagitis NOS (Gastrointestinal disorders) | 6 (11) | 9 (12)
Stomatitis (Gastrointestinal disorders) | 3 (4) | 5 (7)
Toothache (Gastrointestinal disorders) | 3 (3) | 0 (0)
Vomiting NOS (Gastrointestinal disorders) | 17 (37) | 22 (47)
Asthenia (General disorders) | 5 (5) | 5 (9)
Chest discomfort (General disorders) | 2 (2) | 2 (2)
Chest pain (General disorders) | 6 (8) | 4 (5)
Fatigue (General disorders) | 19 (34) | 26 (59)
Influenza like illness (General disorders) | 1 (1) | 2 (3)
Oedema NOS (General disorders) | 2 (2) | 3 (8)
Oedema peripheral (General disorders) | 1 (1) | 4 (6)
Pain NOS (General disorders) | 3 (3) | 2 (3)
Pyrexia (General disorders) | 10 (20) | 14 (22)
Rigors (General disorders) | 3 (4) | 7 (10)
Drug hypersensitivity (Immune system disorders) | 3 (3) | 2 (4)
Candidal infection NOS (Infections and infestations) | 1 (2) | 2 (2)
Lower respiratory tract infection NOS (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia NOS (Infections and infestations) | 4 (4) | 1 (1)
Upper respiratory tract infection NOS (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection NOS (Infections and infestations) | 1 (1) | 2 (2)
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 4 (5) | 5 (5)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 4 (5) | 2 (2)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (2) | 4 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (5)
Blood alkaline phosphatase increased (Investigations) | 2 (5) | 2 (3)
Sputum increased (Investigations) | 2 (3) | 0 (0)
Weight decreased (Investigations) | 5 (5) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 16 (23) | 17 (31)
Dehydration (Metabolism and nutrition disorders) | 5 (6) | 5 (7)
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 3 (3) | 6 (19)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (7)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (5) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (10) | 3 (9)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Local swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 7 (8)
Ataxia (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 3 (5) | 11 (15)
Dysgeusia (Nervous system disorders) | 4 (5) | 7 (7)
Headache (Nervous system disorders) | 7 (10) | 9 (10)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Peripheral neuropathy NOS (Nervous system disorders) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (4) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 4 (4)
Anxiety (Psychiatric disorders) | 0 (0) | 5 (5)
Insomnia (Psychiatric disorders) | 7 (8) | 6 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (24) | 16 (22)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (18) | 16 (26)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (7)
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 14 (16) | 20 (24)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (4)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (5)
Rash NOS (Skin and subcutaneous tissue disorders) | 2 (6) | 3 (3)
Sweating increased (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Hypotension NOS (Vascular disorders) | 4 (5) | 7 (10)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days